CLINICAL TRIAL: NCT06018246
Title: Effects of Different Nutritional Support Modes Based on Nutritional Risk Screening on Postoperative Nutritional Status of Patients With Gastrointestinal Cancer
Brief Title: Nutritional Risk Screening Nutritional Support Gastrointestinal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Huang He, Chief physician of gastrointestinal surgery and Section chief of Medical Services Division, The First Affiliated Hospital of Shanxi Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022HLL003
Record Dates: First submitted 2023-08-15; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 1. Before operation：The patients' dietary intake was assessed by a 24-hour dietary review by a professional dietitian.According to the diet of the patients, the intervention was carried out by a professional nutritionist according to the five-step treatment mode of malnutrition.If the food intake cannot meet 60% of the daily requirement, the previous step of treatment is used, and it is adjusted at any time according to the situation of the patient.
  2. After operation:Same as control group.
  3. Out-of-hospital: Same as before operation.
  4. Strengthening Health Education and psychological intervention:Dietitians need to strengthen health education and communicate with patients during the implementation of nutrition intervention.For patients who actively cooperate with treatment, dietitians can give encouragement.
  5. Exercise Instruction:After the operation, according to the tolerance, the dietitian can instruct the patient to take a certain time walking every day.
  Interventions: Dietary Supplement: Malnutrition five-step treatment model + conventional nutritional intervention
- Control Group (Other): Routine nutrition support in department.Nutritionists will give patients routine parenteral nutrition support via peripheral or central vein 0-48 hours after surgery and then start enteral nutrition support 48-72 hours after surgery.Patients were initially given half of their enteral nutrition and the rest was supplemented with parenteral nutrition.After adaptation, the patient stopped parenteral nutrition and all nutrition came from enteral nutrition.After the patient's gastrointestinal function gradually recovered, the enteral nutrition could gradually decrease.At this time, nutritionists can let the patient eat some light liquid food, but pay attention to eating a small amount of multiple times.After adaptation, patients can gradually transition from liquid diet to semi-liquid diet.We will educate patients and their families about diet and encourage them to eat more high-quality protein-rich foods.
  Interventions: Other: Conventional nutritional intervention

INTERVENTIONS:
Dietary Supplement: Malnutrition five-step treatment model + conventional nutritional intervention — 1. Before operation：Same as arm description.
  2. After operation:Same as control group.
  3. Out-of-hospital: Same as before operation.
  4. Strengthening Health Education and psychological intervention:Dietitians need to strengthen health education and communicate with patients during the implementation of nutrition intervention.For patients who actively cooperate with treatment, dietitians can give encouragement.
  5. Exercise Instruction:After the operation, according to the tolerance, the dietitian can instruct the patient to take a certain time walking every day, gradually increase the patient's muscle endurance and improve the body resistance.
  Arms: Intervention Group
Other: Conventional nutritional intervention — Routine nutrition support in department.Nutritionists will give patients routine parenteral nutrition support via peripheral or central vein 0-48 hours after surgery and then start enteral nutrition support 48-72 hours after surgery.Patients were initially given half of their enteral nutrition and the rest was supplemented with parenteral nutrition.After adaptation, the patient stopped parenteral nutrition and all nutrition came from enteral nutrition.After the patient's gastrointestinal function gradually recovered, the enteral nutrition could gradually decrease.At this time, nutritionists can let the patient eat some light liquid food, but pay attention to eating a small amount of multiple times.After adaptation, patients can gradually transition from liquid diet to semi-liquid diet.We will educate patients and their families about diet and encourage them to eat more high-quality protein-rich foods.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial was to compare the effects of different nutritional support methods based on nutritional risk screening on postoperative nutritional status in patients with gastrointestinal tumors.The main question it aims to answer is that different types of nutrition can improve the nutritional status of patients with different nutritional status;Long-term dietary interventions for patients with poor nutrition can make cancer patients better able to tolerate surgery and chemotherapy and improve their quality of life.The intervention group received nutrition + exercise + psychological intervention upon admission, routine parenteral and enteral nutrition support after operation, and continued nutrition + exercise + psychological intervention after discharge.The control group received routine parenteral nutrition support in the department after surgery, and the patients and their families were given diet education during hospitalization.

DETAILED DESCRIPTION:
Purpose: The investigators conducted nutritional risk screening for patients with gastrointestinal tumors, gave different nutritional support methods to patients with different nutritional status, and analyzed the changes of various nutritional indexes of patients before and after nutritional intervention.

Methods: A total of 302 patients with gastrointestinal tumors admitted to the First Hospital of Shanxi Medical University from July 2021 to June 2023 were selected.All patients underwent nutritional risk screening after admission and were divided into intervention group (NRS2002≥3 and PG=SGA≥4, n=204) and control group (NRS2002 < 3 or PG=SGA < 4 , n=98) according to the screening results.Different nutritional interventions were given to analyze the changes of NRS-2002 and PG-SGA scores between the two groups before and after propensity score matching, and compare the changes of dietary energy, dietary protein, total energy, total protein, body mass index (BMI), fat-free weight, walking time, grip strength and other nutritional indicators (hemoglobin, albumin, prealbumin) between the two groups.The effects of disease type and age on the results were compared by stratified analysis.

ELIGIBILITY:
* Inclusion Criteria:

  1. Age ≥ 18 years；
  2. The first pathological diagnosis was gastric or colorectal cancer and radical resection of malignant tumor was performed；
  3. Conscious, able to read, write and understand the study；
  4. Sign informed consent and participate in this study voluntarily.
* Exclusion Criteria:

  1. Patients with malignant tumors at other sites；
  2. Patients undergoing neoadjuvant chemotherapy before surgery；
  3. Anastomotic fistula, anastomotic obstruction, gastroparesis and other serious complications occurred after operation；
  4. There are mental disorders, psychological disorders；
  5. Patients who did not cooperate to complete the full intervention or follow-up records were missing；
  6. Patients with missing baseline data and nutritional risk screening results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Nutritional risk screening 2002 | baseline and through study completion, an average of 1 year
  Nutritional risk screening scale：The maximum score of NRS2002 is 7 points and the minimum score is 0 points. A score of NRS2002≥3 indicates the presence of nutritional risk, and nutritional support programs should be developed in combination with clinical practice. A score of NRS2002 < 3 indicates no nutritional risk, and a review is performed 1 week later.
Patient-generated subjective nutrition assessment | baseline and through study completion, an average of 1 year
  Nutritional risk screening scale：0-1 score, no intervention is required at this time, regular regular nutritional status score. 2 to 3 points, the nutritionist, nurse or clinician to educate the patient and family, and appropriate drug intervention for symptoms and laboratory tests. 4-8 points, requiring nutritional intervention and symptomatic treatment. A score of ≥9 indicates an urgent need for symptomatic treatment and appropriate nutrient support.

SECONDARY OUTCOMES:
Dietary energy intake | baseline 、7 days after admission、1 month after admission、2 month after admission、4 month after admission and through study completion, an average of 1 year
  The 24-hour dietary review method was used to investigate the diet of the patients in the first 24 hours, and all the foods were converted into the energy value of the foods, and the dietary energy intake of the patients was calculated by adding.
Dietary protein intake | baseline 、7 days after admission、1 month after admission、2 month after admission、4 month after admission and through study completion, an average of 1 year
  The 24-hour dietary review method was used to investigate the diet of the patients in the first 24 hours, and the protein amount provided by each food was recorded, and the dietary protein intake of the patients was calculated by adding.
Nutrient energy intake | baseline 、7 days after admission、1 month after admission、2 month after admission、4 month after admission and through study completion, an average of 1 year
  The nutritional energy provided by oral nutrition, enteral nutrition and parenteral nutrition was recorded through inquiry and inquiry of nursing records.
Nutrient protein intake | baseline 、7 days after admission、1 month after admission、2 month after admission、4 month after admission and through study completion, an average of 1 year
  The nutritional proteins provided by oral nutrition, enteral nutrition and parenteral nutrition were recorded through inquiry and inquiry of nursing records.
Prealbumin | baseline 、7 days after admission、1 month after admission、2 month after admission、4 month after admission and through study completion, an average of 1 year
  Laboratory indicators on nutrition
Albumin | baseline 、7 days after admission、1 month after admission、2 month after admission、4 month after admission and through study completion, an average of 1 year
  Laboratory indicators on nutrition
Hemoglobin | baseline 、7 days after admission、1 month after admission、2 month after admission、4 month after admission and through study completion, an average of 1 year
  Laboratory indicators on nutrition
BMI | baseline 、7 days after admission、1 month after admission、2 month after admission、4 month after admission and through study completion, an average of 1 year
  Dietitians use a body fat scale to measure a patient's weight.When measuring the patient's weight, the body fat scale should be placed on a horizontal, firm floor.The patient takes off shoes and socks and wears light clothes.The patient then stood on the scale, keeping his body naturally upright.The patient's arms should be naturally drooped and relaxed at the sides of the body.Each weight measurement should be set at the same time.The dietitian uses a height meter to measure the patient's height.Weight and height will be combined to report BMI in kg/m^2.
Fat-free body weight | baseline 、7 days after admission、1 month after admission、2 month after admission、4 month after admission and through study completion, an average of 1 year
  Dietitians use a body fat scale to measure a patient's fattened weight.When measuring the patient's weight without fat, the body fat scale should be placed on a level, firm floor.The patient takes off shoes and socks and wears light clothes.The patient then stood on the scale, keeping his body naturally upright.The patient's arms should be naturally drooped and relaxed at the sides of the body.The weight loss should be measured at the same time each time.
Grip strength | baseline 、7 days after admission、1 month after admission、2 month after admission、4 month after admission and through study completion, an average of 1 year
  A dietitian uses a grip dynamometer to measure a patient's grip strength.When grip strength is measured, the patient's hands naturally droop and no other hand movements can be seen.Dietitians advise patients to measure their grip strength as best they can.The patient is tested on both hands, usually three times with each hand, and an average is taken.
Walking time | baseline 、7 days after admission、1 month after admission、2 month after admission、4 month after admission and through study completion, an average of 1 year
  The patients were asked about their daily walking time.

OTHER OUTCOMES:
Adverse reaction | baseline 、7 days after admission、1 month after admission、2 month after admission、4 month after admission and through study completion, an average of 1 year
  After the clinician and dietitian judge the occurrence of adverse reactions, the types of adverse reactions are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, doctor's degree, Study Director — The First Affiliated Hospital of Shanxi Medical University
Locations (1):
- Huang He, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No